CLINICAL TRIAL: NCT05603793
Title: YoUng Adolescents' behaViour, musculoskeletAl heAlth, Growth & Nutrition
Acronym: YUVAAN
Status: Active, not recruiting | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Deputy director, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: YUVAAN
Record Dates: First submitted 2022-10-10; First posted 2022-11-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Arrest of Bone Development or Growth; Constitutional Delay of Growth and Puberty; Malnutrition, Child; Gestational Diabetes; Muscle Tone Abnormalities; Anemia
Keywords: adolescent; growth; malnutrition; cycle of nutrition; cohort
MeSH Terms: conditions — Child Nutrition Disorders; Diabetes, Gestational; Anemia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Knowledge, Attitude & Practices — The objective the of the KAP intervention is to explore key aspects related to child health and nutrition to better understand the community's knowledge, perception and practices. In addition to child health, we are also tracking the transition of health from urban to rural areas in terms of the prevalence of adult non-communicable diseases.

SUMMARY:
More children will survive to adulthood today than at any other point in human history, as evidenced by the proportion of live births and absolute numbers. The present generation of young people who have lived to the age of five will reach adulthood around 2030 and will be the generation of the Sustainable Development Goals (SDGs). These children's health and nutrition as they grow from 5 to 19 years will have permanent ramifications on the development of the coming generation.

The Comprehensive National Nutrition Survey was conducted between 2016 and 2018, indicating unacceptably high levels of malnutrition among Indian children and adolescents. It was discovered that one out of every five children aged 5 to 9 was stunted, indicating they were malnourished for their age. Undernourished girls are more likely to become short-statured mothers, giving birth to low-birth-weight and stunted newborns who are more prone to disease and linear growth failure. Evidence suggests that maternal short stature (less than 150 cm) predicts childhood growth failure and increases the risk of having a stunted baby by two years. The common genetic background and environmental influences that affect the mother during her early childhood and adolescence play a substantial role in the relationship between maternal stature and the linear growth of the child. This causes a cycle of undernutrition and poor growth that continues through generations and impacts the offspring's growth.

Adolescence is a key period of physical and social development when the physiological, mental, and behavioural underpinnings of long-term health are established. The development of critical bone mass is crucial during this time because it lays the foundation for preserving bone mineral integrity later in life. During adolescence, over 40% of peak bone mass is achieved. Changes in body composition are also seen during early adolescence. These physiological processes are both nutritionally sensitive and predictive of their future health. Adolescent behaviour is also linked to 33 percent of sickness and 60 percent of premature deaths in adulthood. Because adolescence is also a critical period for the development of the ability to make independent decisions, follow them through, and achieve goals- enabling healthy social networks, is critical. This includes Social and Behavioural Change Communications, which can assist early adolescents create lifetime behaviour patterns, such as good nutrition and physical exercise choices.

Investing in adolescent health and well-being pays off in three ways: during their adolescence, in their adulthood, and for their future offspring generations. Thus, young adolescence provides a "window of opportunity" for children to improve their nutritional health and outcomes.

Therefore, this cohort aims to explore the trajectories of growth (including anthropometric measures, bone mass, and muscle mass and function) among rural young adolescents and its association with intergenerational nutritional status through a longitudinal study.

A greater understanding of growth trajectories set in a longitudinal study would aid in the discovery of particular variables that influence the timing of young adolescents' growth and the factors associated with intergenerational nutritional status.

DETAILED DESCRIPTION:
Aims and Objectives

Aim:

This cohort aims to study the adolescent growth trajectory of girls and boys aged 8 to 10 years from rural Maharashtra. The impact of these indicators on their future offspring size will be studied by following the adolescent cohort and assessing their intergenerational nutritional status till their first offspring is 5 years old.

Objectives:

1. To study trajectories of growth (height/ weight/ body mass index/ growth velocity) among young adolescents aged 8 to 10 years in rural areas of Maharashtra.
2. To longitudinally study the acquisition of bone mass, muscle mass, and function in young adolescents aged 8 to 10 years in rural areas of Maharashtra.
3. To study the association of intergenerational nutritional status among young adolescents in comparison with their parent's height and future offspring size and body composition.
4. To strengthen Social and Behavioural Change Communication (SBCC) strategies that impact the nutritional status of young adolescents and their parents by exploring and improving their Knowledge, Attitude, and Practices.

Proposal The adolescent cohort study is a longitudinal community-based study of pre-adolescents of age between 8 to 10 years.

Primary Participants: A cohort of pre-adolescents aged 8 to 10 years, who fulfil the inclusion criteria will be enrolled from 8 villages.

Secondary Participants: The parents of the included young adolescents will also be enrolled in the cohort, to study intergenerational effects.

The enrollment period will be set for two years.

Inclusion Age between 8 and 10 years during the period of enrollment Children with both biological parents (mother and father) present during the period of enrollment Apparently healthy children

Exclusion Any chronic untreated/ progressive condition that would adversely affect the growth, bone and/or muscle health of the participant Migrant families and temporary residents as defined by the Census of India (as defined by the Office of the Registrar General & Census Commissioner, India Ministry of Home Affairs, 2022) Refusal to give informed consent and/or parental assent

Geographic location and village screening The study covers 8 villages from Shirur, Block of Pune district in Maharashtra, India, which fulfil the inclusion criteria for being 'rural' as defined by the Census of India (as defined by the Census of India, 2021).

The population is homogeneous in living conditions, socioeconomic status, and dietary habits. Most people are engaged in agriculture and have a low migration rate, which makes it an optimal setting for conducting cohort studies.

Since our study aims to find the association between intergenerational nutritional status and growth in three generations, the study will extend for years. For such long-duration investigations, it was important to select study cohorts that are not likely to migrate, are cooperative and are likely to be so throughout the study, and most importantly, easily accessible to the investigators so that the expense and efforts are kept within reasonable limits.

Peripheral quantitative computed tomography (pQCT), and Dual-energy X-ray absorptiometry (DXA) scanners are not available in most healthcare centres in rural India. This limitation in availability made the study be set in villages near the HCJMRI health centre, Ranjangaon where the units already exist. Since Ranjangaon is an industrial area, an increase in-migrant workers were seen, hence it was excluded.

The cost of such a study, as well as the need to ensure its operation over 20 years, puts it beyond the capability of researchers. Thus, if such a study is to be carried out, it is evident that it will need the help of local community health agencies. Thus, villages with uncooperative stakeholders (such as healthcare staff, community leaders, and so on) were omitted.

It is not possible to conduct measurements in multiple regions at the same time due to the high cost of examination and follow-up. As a result, it was decided that the study should be divided into two groups of four villages (n=8) clustered together. Two sets were chosen if cohort matching studies were required in the future.

From an administrative aspect, office facilities had to be secured, as well as one field staff for each community. On either side of the National Highway (which served as a marker for demarcation), four villages that met the inclusion criteria were chosen. A residential structure in the middle of the four villages was converted into office space. Data is collected twice a week, after which it is monitored, processed, and sent to the main office by staff once a week.

Sampling

The investigators are recruiting study subjects from 8 villages in Shirur taluka (In the rural areas the smallest area of habitation, viz., the village generally follows the limits of a revenue village that is recognized by the normal district administration):

Group A: Vaghale, Varude, Ganegaon Khalsa and Pimpale Khalsa Group B: Nimgaon Mhalungi, Karde, Bhambarde, Karanjawane A three-stage design (Taluka-Village-Household) was used. Stratification was done based on the geographical and gender-wise distribution to provide a proportionate minimum sample of young adolescents aged 8 to 10 years that was truly representative of the population under study.

Training Before beginning fieldwork, all field personnel had received extensive training. The training program included standardized data collection, management, and processing seminars. Print and digital media aids were also used in the training (e.g., standardized videos dubbed in local languages, and show cards). Field workers were also taught how to create rapport, communicate effectively, make appropriate referrals, initiate community development activities, and administer first aid. After the training program, all trainees were evaluated. Training is a continuous process that will include refresher sessions (at least 6monthly) on the field.

Execution of fieldwork

Pre-field activities Pre-field activities began by seeking and obtaining approval from health authorities in the taluka. Permission was then obtained from the panchayat head/village elder to be able to enter the village to conduct the study.

Pre-field activities also included inventory counts (medical supplies, instruments, stationery, etc.) and equipment calibration.

Preliminary Data The investigators had previously conducted studies across these areas to determine the health status of the people living in and around these villages. Previous studies conducted by the team provided preliminary data to recognize the gaps. Studies were conducted to identify the relationships between parental body size and maternal gestational weight gain with their offspring size at birth as well as adolescent growth status, muscle mass, and bone strength.

The preliminary work from 2020 in areas around Ranjangaon enrolled 124 pregnant women (<12 weeks). The cohort of pregnant women and their spouses showed a positive correlation (p≤ 0.05) between paternal height and the birth weight of their offspring, suggesting that the impact of intergenerational nutritional status could be explained by genetic factors.

Growth, bone health, and muscle function were also found to be lower than reference values among young adolescents in rural parts of India.

Field activities

Ethical Clearance & Consent Before the start of the study, the senior staff and researchers of HCJMRI met the village authorities and community leaders to explain the aims of the study and to ensure people's interest in participation and compliance with follow-up assessments. The PI is asked by the field investigators for each family's eligibility to take part in the study. Approval for the study has been obtained from the institutional ethics committee.

Participant Information Sheet The participant information sheet (PIS) is used to explain the purpose and importance of the study and the participant's involvement. The PIS is available to the target audience in their local language (Marathi). A copy of the PIS is available in English for the PI.

Informed Consent The research assistant enters the eligible participant's initials and date of birth into an 'Initial table for Recruiting' spreadsheet and assigns an enrolment number. There is one spreadsheet per village. A participation information sheet (PIS) and consent form is administered in the local language (Marathi) and signatures of the participants (and participants' parents) are sought. In case of illiterate individuals, the PIS is narrated in Marathi, and a thumb impression (witnessed by a person unrelated to the study) is taken. Sufficient time is allocated to participants and their parents to ask questions and have them answered to their satisfaction. For children (8-10 years), written parental consent is obtained with assent from the child. All forms are signed by PI/Co-PI.

Components of the data collection form The questionnaire is structured, and close-ended with sections on data collection for household data, fathers data, mothers data and young adolescents data. After the primary participant has their offspring, an extra section will be added to collect offspring data as well.

Household data includes socio-demographics like education and occupation of the head, the list of family members present in one household and the monthly family income. Participants' medical history, clinical assessment, sunlight exposure, physical activity and dietary intake is assessed using validated questionnaires. All enrolled participants are mapped for future reference, post receiving their consent.

Anthropometric measurements include height, weight, body composition and MUAC for young adolescents.

Biochemical markers include the parents' Haemoglobin and Blood Sugar Levels (BSL).

Haemoglobin, BSL, and indicators of bone metabolism and growth modulators- Calcium Phosphate, Alkaline Phosphatase, Parathyroid Hormone (PTH), vitamin D, Serum Creatinine and Luteinizing Hormone (LH) is tested in young adolescents. Serum calcium, phosphorus, 25-hydroxyvitamin D, and parathyroid hormone are common calcium homeostasis indicators, however, they do not directly reflect bone turnover. As a result, the investigators combine them with comprehensive medical, menstrual (for girls), and family history; a thorough system assessment; and a directed objective examination, which includes BMI calculation and skeletal bone age.

Further insight into bone accrual is obtained by measuring bone acquisition and bone mineral density (BMD) using non-invasive bone evaluation techniques through DXA and pQCT. Muscle function and muscle strength is measured through Jumping Mechanography and a hand dynamometer.

The anthropometric, physical activity, sunlight exposure and dietary intake details is collected biannually. The muscle, bone and blood investigations is performed annually among young adolescents and biyearly in their parents.

Training of field workers

Each village is represented by one field worker. The field workers are village residents, between the ages of 30 and 45. They are taught how to communicate effectively and how to lead others. With formal schooling up to eighth grade, they are literate enough to administer the data collection form.

Field personnel conduct a baseline door-to-door survey to obtain willingness to participate and shortlist eligible participants for the study. Field personnel are carefully selected based on their understanding of the language and population. They trained for two weeks by senior investigators in the use of instruments to assure uniformity of data. Intra and inter-observer variability of measurements are assessed at the beginning of the study and periodically every 6 months. It is noticed that some participants in the family will be missed by the field worker at their first assessment after enrollment. This is largely due to other commitments by the participant on the day of their attendance. In such cases, the participant is visited again by the field worker.

Standard Operating Procedures (SOPs) SOPs have been established and distributed to the research and field teams, with specific instructions on how to record investigations, processes, and activities. The SOPs specify the methods and systems that will be used to ensure that field and research duties are completed in compliance with institutional norms.

Pretesting and piloting of data collection items The data collection form was pretested by researchers and clinicians from the fields of paediatrics and public health. An individual assessment of each item was provided and rated on a Likert scale. This was done to collect the experts' opinions and judgement of how well the questionnaire reflected the construct, which the investigators intended to measure in a community-based setting.

Piloting was done on families of 10 young adolescents belonging to Ganegaon Khalsa and Karanjawne, who fit the inclusion criteria. Data collection for one participant took 30-40 minutes, and for one family of 3 members took 1 hour and 40 minutes, including the measurements and blood sample collection. Piloting was also necessary since the questionnaire was administered through field workers in the local language. The pilot test helped us identify inconsistencies and irregularities in the language and accessibility issues within the survey instrument. After piloting, the major issues with questions, measurement, and design which were apparent were resolved.

Post-field activities

Data quality and management The data was assessed on several dimensions, such as key variable accuracy, completeness of all required attributes, data consistency, timeliness, and so on. Location data with geographic coordinates was also mapped for individual households.

Project Implementation Every six months, all enrolled households will be visited, and data on anthropometric parameters, migrations, updated contact numbers, pubertal status, and self-reported common illnesses, etc will be gathered. Every death will be subjected to a verbal autopsy (VA).

Community Engagement and maintenance of cohort The field investigators will be in constant touch with the families through social media and Whatsapp. Whatsapp groups will also help in referrals and record events that affect the cohort like migration, marriages, absenteeism due to acute illnesses, etc.

SWOT Analysis

Strengths Previous health camps conducted Existing relationships with community leaders Experienced project team

Opportunities Connectivity with participants due to increased internet usage Geographic coverage of the study: heterogeneous population Lesser penetration by other healthcare organisations

Weaknesses Reluctance from family members Limited capacity in data storage and monitoring

Threats Bad communication networks Migration of participants Risks to the security of collected data

Agency Profile

Hirabai Cowasji Jehangir Medical Research Institute (HCJMRI) was founded in 1995 with the objective of contributing to Scientific Research and improving the quality of life of humans. HCJMRI is a sister concern of the Jehangir Hospital, Pune and is situated on the premises of the Hospital.

HCJMRI is recognized by the Directorate of Scientific and Industrial Research (DSIR), Government of India as a centre for multi-disciplinary research in various branches of research and holds a prestigious certificate which allows maximum tax exemption to donors (35 I ii).

Project Interventions

Expected Outcomes

1. The study will help track growth and bone acquisition trajectories in rural adolescents.
2. The study will throw light on intergenerational malnutrition and its associations.
3. The study will help in identifying modifiable factors associated with malnutrition.
4. Data collected in the study as well as results will be shared with stakeholders and policymakers.
5. Due to the nature of the study, it will help in health and nutrition awareness in the community
6. Results of the study will be shared through scientific publications and lay press
7. Data from the study will be available for secondary data analysis upon reasonable request.

Sustainability of the Project The inclusion of adolescent health in the UN Secretary-Global General's Strategy on Women's and Children's Health, as well as targets directly related to adolescent health in the post-2015 Sustainable Development Goals agenda, represents a once-in-a-lifetime opportunity to accelerate efforts to adopt policies for young adolescents. Countries can guarantee that young adolescents contribute fully to their society and acquire the judgement, values, behaviours, and resilience they need by being safe and healthy. This can be done through undertaking research projects concentrating on their health and development, particularly in lower and middle-income settings. As a result, this healthy generation will nurture the next, allowing them to effectively participate in a constantly changing globalised world.

Many countries may profit from rapid economic growth associated with the demographic dividend if today's growing young adults are combined with low fertility, increased health, nutrition, and education.

Way Forward Renewing investments in adolescent health will make significant contributions to the progressive realisation of children's rights under the Convention on the Rights of the Child and the Convention on the Elimination of All Forms of Discrimination Against Women, as well as to the achievement of Sustainable Development Goals 3, 5, and 10.

ELIGIBILITY:
Inclusion

* Age between 8 and 10 years during the period of enrollment
* Children with both biological parents (mother and father) present during the period of enrollment
* Apparently healthy children

Exclusion

* Any chronic untreated/ progressive condition that would adversely affect growth, bone and/or muscle health of the participant
* Migrant families and temporary residents as defined by Census of India (Office of the Registrar General & Census Commissioner, India Ministry of Home Affairs, 2022)
* Refusal to give informed consent and/or parental assent

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population is homogeneous in living conditions, socioeconomic status, and dietary habits. Most people are engaged in agriculture and have a low migration rate, which makes it an optimal setting for conducting cohort studies.
  Since our study aims to find the association between intergenerational nutritional status and growth in three generations, the study will extend to years. For such long-duration investigations, it was important to select study cohorts that are not likely to migrate, are cooperative and are likely to be so throughout the duration of the study, and most importantly, easily accessible to the investigator so that the expense and efforts are kept within reasonable limits (Banerjee & Chaudhury, 2010).
Sampling Method: Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2047-09-25 (Estimated); Study Completion 2050-09-25 (Estimated)

PRIMARY OUTCOMES:
Wasting | From date of enrolment, until study completion, assessed every 6 months
  Wasting measured as < -2 Weight-for-height z-score
Stunting | From date of enrolment, until study completion, assessed every 6 months
  Stunting measured as < -2 Height-for-age z-score

SECONDARY OUTCOMES:
Body mass and composition | From date of enrolment, until study completion, assessed every 6 months
  Fat percentage measured through the bioelectrical impedance analysis (BIA) method (Tanita Body Composition Analyzer (Model BC-420MA)
Dynamic muscle function | From date of enrolment, until study completion, assessed every 1 year
  Measured using Leonardo Mechanography GRFP version 4.4, Novotec expressed in standard deviations above and below the average
Bone mineral density (BMD) | From date of enrolment, until study completion, assessed every 1 year
  Using dual energy X-ray absorptiometry (Lunar iDXA) expressed in standard deviations above and below the average
Bone volumetric density | From date of enrolment, until study completion, assessed every 1 year
  Using peripheral quantitative computed tomography (pQCT, Stratec XCT 2000) expressed in standard deviations above and below the average
Bone age | From date of enrolment, until study completion, assessed every 6 months
  To estimate the maturity of the child's skeletal system by taking an X-ray of the left wrist. The bones on the X-ray image are compared with X-ray images in a standard atlas of bone development. The atlas is based on data from many other kids of the same gender and age. The bone age (also called the skeletal age) is measured in years.

OTHER OUTCOMES:
Household Dietary Diversity Scale (HDDS) | From date of enrolment, until study completion, assessed every 6 months
  The HDDS reflects household access to food variation and is a count of the food groups consumed over a given reference period. The value of this variable will range from 0 to 12 and represents the total number of food groups consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha V Khadilkar, MD, Principal Investigator — HCJMRI
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miriam D, Mandlik R, Patwardhan V, Ladkat D, Khadilkar V, Kajale N, More C, Gondhalekar K, Bhawra J, Katapally TR, Khadilkar AV. An observational, multigenerational platform for health systems and population health interventions to minimise intergenerational transmission of non-communicable diseases in India: the YUVAAN cohort study protocol. BMJ Public Health. 2025 Feb 6;3(1):e001741. doi: 10.1136/bmjph-2024-001741. eCollection 2025. PMID 40017955
- See also: Cardiovascular and metabolic consequences of obesity. — https://www.frontiersin.org/articles/10.3389/fphys.2015.00032/full
- See also: Maternal and child undernutrition and overweight in low-income & middle-income countries — https://pubmed.ncbi.nlm.nih.gov/23746772/
- See also: Prevalence and factors associated with anemia in 6-18 years urban and rural Indian children and adolescents: A multicenter study. — https://mansapublishers.com/index.php/ijch/article/view/2404
- See also: Determinants of muscle power and force as assessed by Jumping Mechanography in rural Indian children. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8919658/